CLINICAL TRIAL: NCT01285154
Title: Modified Triple Osteotomy for Acetabular Dysplasia - A Modified Technique for Better Femoral Head Medialization and Coverage
Brief Title: Modified Triple Osteotomy for Acetabular Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Li, Yi-Chen, National Taiwan University Hospital
Other Study IDs: 201012045RC
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-01

CONDITIONS: Sharp Angle; Center Edge Angle; Femoral Head Extrusion Index; Center Head Distance Discrepancy
Keywords: Hip dysplasia; Triple Osteotomy; Femoral Head Coverage; Femoral Head Medialization
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traditional Steel Triple Osteotomy: Traditional technique
- Modified Triple Osteotomy: Modified technique

SUMMARY:
Steel triple innominate osteotomy was designed for dysplastic hip in adolescents and young adults with three incisions to increase the coverage; however the amount of correction remained questionable due to ligamentous attachments that hinder the rotation. The investigators modified the technique with two anterior incisions and ramus cuts close to inferior acetabulum. The purpose of this study is to compare these two techniques in femoral head coverage

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic acetabular dysplasia in adolescent or young adult
2. Closed triradiate cartilage
3. Minor coxarthrosis with Tonnis grades at 1 or 2

Exclusion Criteria:

1. High subluxation or complete dislocation of the hip joint
2. Severe osteoarthrosis
3. Combined with proximal femoral osteotomy that changed the femoral neck shaft angle (such as varus or valgus osteotomy)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Young adults and adolescents underwent triple innominate osteotomy for symptomatic acetabular dysplasia in our institution
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Li, M.D., Study Chair — National Taiwan University Hospital, Department of Orthopaedic Surgery
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan